CLINICAL TRIAL: NCT04616482
Title: Supporting and Enabling Physicians to Deliver Personalized Therapeutic Nutrition Using an Online Technology Platform
Brief Title: Therapeutic Nutrition With Technology in Primary Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Associate Professor, University of British Columbia
Other Study IDs: H19-00316
Record Dates: First submitted 2020-10-08; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Diet Modification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Digital therapeutic carbohydrate restriction (TCR) program: The intervention involves 12 weeks of online/app-based behaviour change coaching. Each week the participant focuses on a different aspect of healthy eating habits designed to cut sugar and refined carbohydrates while encouraging and providing resources for lower-carbohydrate food options. Education is done through short videos and information sheets. Participants set goals and complete worksheets/tasks based on their individual goals.
  Interventions: Behavioral: Digital therapeutic carbohydrate restriction (TCR) program

INTERVENTIONS:
Behavioral: Digital therapeutic carbohydrate restriction (TCR) program — A 12-week, personalized, online program to teach and coach patients about therapeutic carbohydrate restriction as for obesity and/or T2D (or risk of T2D). The program is intended to enhance the usual clinical care provided for patients.

SUMMARY:
Low-carbohydrate diets (less than approximately 130 grams per day) are emerging as an efficacious treatment option with several studies supporting weight loss and remission of type 2 diabetes. Many physicians are now implementing this strategy but the time it takes to educate patients on nutrition is a barrier. The research team is working with physicians to develop a solution whereby the nutrition education and intervention is delivered via mobile/online technology (i.e., an app). This study will test whether it is feasible and efficacious for physicians to recommend this app to their patients with obesity and type 2 diabetes to help them lose weight and improve their condition.

DETAILED DESCRIPTION:
The study is a non-experimental feasibility study to explore the acceptability, practicality and demand for the use of a 12-week, personalized, online program to teach and coach patients about therapeutic carbohydrate restriction for individuals with obesity and/or at risk for type 2 diabetes/with type 2 diabetes. The program is intended to enhance the usual clinical care provided for patients with these conditions and will allow for physicians to monitor patient progress through the program. Both physician and patient perspectives will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese (BMI >25 kg/m2)
* At risk for T2D as deemed by physician
* Diagnosed with T2D
* Able to read and speak English (in order to communicate with the technology platform/app
* Over the age of 18

Exclusion Criteria:

* Unable to read or speak English (due to the app being provided in English)
* Unable to access a computer or mobile phone that has access to the internet.
* Currently compliant with a very low carbohydrate ketogenic diet or very low calorie commercial weight loss program
* Planning to change doctors in the next 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with obesity, at risk for type 2 diabetes or diagnosed with type 2 diabetes interested in therapeutic carbohydrate restriction for management of their condition.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
The percentage of eligible patients who receive prescriptions to access the online TCR program | through study completion, an average of 9 months
  Assessed through the number of voucher cards handed-out over physician documentation of eligible patient visits over the study period.

SECONDARY OUTCOMES:
Present descriptive characteristics of patients who get prescriptions to access the online TCR program | through study completion, an average of 9 months
  Assessed through program intake collected through the online program (e.g. age, sex, weight, HbA1c, chronic condition, health goals)
The percentage of patients who receive a prescription for TCR program that sign up and start | through study completion, an average of 9 months
  Assessed through the number of voucher cards redeemed on the online program over the number of voucher cards handed-out by physicians.
Program drop-out as assessed by the number of patients who sign up for and start the TCR program and the number of patients who complete the full program. | Pre-program (month 0) to post-program (6 months)
  Assessed through the number of patients enrolled in the program and the number of patients who complete the program through program tracking.
Program impact assessed through changes in weight from pre-program to post-program. | Pre-program (month 0) to post-program (6 months)
  For patients who complete the program, the change in weight from program sign-up to program completion.
Program impact assessed through change in HbA1c from pre-program to post-program. | Pre-program (month 0) to post-program (6 months)
  For patients who complete the program, the change in HbA1c from program sign-up to program completion.
Program impact assessed through changes in medications from pre-program to post-program. | Pre-program (month 0) to post-program (6 months)
  For patients who complete the program, the change in medications from program sign-up to program completion.

OTHER OUTCOMES:
Qualitative patient feedback on program acceptability | Post-program (6 months)
  Qualitative semi-structured interviews with patients collecting program feedback on their experiences in the program, specifically asking about the acceptability of the program. Acceptability will be assessed through the audio-recorded responses to semi-structured interview questions, subsequently transcribed and coded using content analysis.
Qualitative patient feedback on program practicality | Post-program (6 months)
  Qualitative semi-structured interviews with patients collecting program feedback on their experiences in the program, specifically asking about the practicality of the program. Practicality will be assessed through the audio-recorded responses to semi-structured interview questions, subsequently transcribed and coded using content analysis.
Qualitative patient feedback on program satisfaction | Post-program (6 months)
  Qualitative semi-structured interviews with patients collecting program feedback on their experiences in the program, specifically asking about their satisfaction of the program. Satisfaction will be assessed through the audio-recorded responses to semi-structured interview questions, subsequently transcribed and coded using content analysis.
Qualitative physician feedback on program acceptability | through study completion, an average of 9 months
  Qualitative semi-structured interviews with physicians collecting feedback on their experiences in the program, specifically asking about the acceptability of the program within their daily physician practice. Acceptability will be assessed through the audio-recorded responses to semi-structured interview questions, subsequently transcribed and coded using content analysis.
Qualitative physician feedback on program practicality | through study completion, an average of 9 months
  Qualitative semi-structured interviews with physicians collecting feedback on their experiences in the program, specifically asking about the practicality of the program within their daily physician practice. Practicality will be assessed through the audio-recorded responses to semi-structured interview questions, subsequently transcribed and coded using content analysis.
Qualitative physician feedback on program satisfaction | through study completion, an average of 9 months
  Qualitative semi-structured interviews with physicians collecting feedback on their experiences in the program, specifically asking about the satisfaction of the program within their daily physician practice. Satisfaction will be assessed through the audio-recorded responses to semi-structured interview questions, subsequently transcribed and coded using content analysis.
Characteristics of individuals who drop-out of program | through study completion, an average of 9 months
  Provide descriptive statistics (e.g. age, sex, weight, HbA1c, chronic condition, health goals) of individuals who drop-out after enrolling in the program and prior to program completion.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon Little, PhD, Principal Investigator — The University of British Columbia, Okanagan Campus
Locations (1):
- University of British Columbia Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No